CLINICAL TRIAL: NCT02439411
Title: Retrospective Analysis of Dabrafenib +/- Trametinib Compassionate Use Experience in Spain
Acronym: DEIS
Status: Completed | Type: Observational
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: GEM1401
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Malignant Melanoma Stage IV; Malignant Melanoma Stage IIIc
MeSH Terms: conditions — Melanoma | interventions — trametinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Dabrafenib
- Dabrafenib plus Trametinib: Patients treated with Dabrafenib plus Trametinib
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: Trametinib
  Groups: Dabrafenib plus Trametinib

SUMMARY:
The purpose of this study is to analyze whether Dabrafenib +/- Trametinib are effective in overall survival, response rates and toxicity in both programs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received at least one dose of dabrafenib or combination with trametinib as part of a compassionate use for the treatment of metastatic melanoma, with deadline the start of treatment the April 30, 2014.

Exclusion Criteria:

* Patients with a history not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastasic melanoma patients treated with Dabrafenib +/- Trametinib in compassionate use.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Best Overall Response | Up to 18 months
  Participants will be followed for the duration of hospital stay, an expected average of 18 months.
Adverse Event Rates | Participants will be followed for the duration of hospital stay, an expected average of 18 months.
  Percentage of patients developing an Adverse Event through follow-up

SECONDARY OUTCOMES:
Overall Survival | Participants will be followed for the duration of hospital stay, an expected average of 18 months.
  Number of patients alive at the end of the follow-up period and median time between start of treatment and death.
Resectability of tumor | Participants will be followed for the duration of hospital stay, an expected average of 18 months.
  Proportion of patients whom tumor was resectable
Adherence to treatment | Participants will be followed for the duration of hospital stay, an expected average of 18 months.
  Proportion of patients who comply with treatment as prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Martín Algarra, M.D., Ph.D., Study Chair — Clinica Universidad de Navarra
Locations (29):
- Spain (29):
  - Complejo Hospitalario Torrecárdenas, Almería, Almería
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Instituto Catalán de Oncología Badalona/Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Instituto Catalán de Oncología L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Corporació Sanitaria Parc Taulí de Sabadell, Sabadell, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Onkologikoa Fundazioa, Donostia / San Sebastian, Guipúzcoa
  - Complejo Hospitalario Universitario Insular de Canarias, Las Palmas de Gran Canaria, Las Palmas
  - Clínica Universidad Navarra, Pamplona, Navarre
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Instituto Catalán de Oncología Girona/Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitaria La Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Valme, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martin Algarra S, Soriano V, Fernandez-Morales L, Berciano-Guerrero MA, Mujika K, Manzano JL, Puertolas Hernandez T, Soria A, Rodriguez-Abreu D, Espinosa Arranz E, Medina Martinez J, Marquez-Rodas I, Rubio-Casadevall J, Ortega ME, Jurado Garcia JM, Lecumberri Biurrun MJ, Palacio I, Rodriguez de la Borbolla Artacho M, Altozano JP, Castellon Rubio VE, Garcia A, Luna P, Ballesteros A, Fernandez O, Lopez Martin JA, Berrocal A, Arance A. Dabrafenib plus trametinib for compassionate use in metastatic melanoma: A STROBE-compliant retrospective observational postauthorization study. Medicine (Baltimore). 2017 Dec;96(52):e9523. doi: 10.1097/MD.0000000000009523. PMID 29384960